CLINICAL TRIAL: NCT02305537
Title: Building an Outcomes Assessment Infrastructure to Assess Youth in the McLean Anxiety Mastery Program at McLean Hospital
Brief Title: Building an Outcomes Assessment Infrastructure to Assess Anxiety Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Sperling, Jacqueline,Ph.D., Associate Program Director of the McLean Anxiety Mastery Program, Mclean Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014P000353
Record Dates: First submitted 2014-11-14; First posted 2014-12-02 (Estimated); Last update posted 2025-10-20 (Actual); Status verified 2023-03

CONDITIONS: Social Anxiety Disorder; Specific Phobia; Separation Anxiety Disorder; Panic Disorder; Agoraphobia; Obsessive-Compulsive Disorder
MeSH Terms: conditions — Phobia, Social; Phobia, Specific; Anxiety, Separation; Panic Disorder; Agoraphobia; Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Cognitive-Behavioral Therapy) (Experimental): Participants in the McLean Anxiety Mastery Program
  Interventions: Behavioral: McLean Anxiety Mastery Program
- Waitlist (No Intervention): Participants on the waitlist for the McLean Anxiety Mastery Program

INTERVENTIONS:
Behavioral: McLean Anxiety Mastery Program — Cognitive-Behavioral Therapy with Exposure and Response Prevention
  Arms: Treatment (Cognitive-Behavioral Therapy)

SUMMARY:
The collection of patient self-report and diagnostic data will allow us to examine the efficacy of the treatment delivered in the McLean Anxiety Mastery Program. Using data gathered through routine clinical care, the investigators seek to explore whether patients in treatment show improvements from admission to discharge, compared to patients on the waitlist, and whether these gains are maintained three months post-discharge. The following are included as examples of some of the study's hypotheses.

DETAILED DESCRIPTION:
The study population will involve all assenting/consenting patients, both male and female, admitted to the McLean Anxiety Mastery Program at McLean Hospital. This program provides intensive group-based treatment for anxious youth (aged 6-19). Patients in the McLean Anxiety Mastery Program participate in a minimum of four weeks of treatment and attend the program for four days per week. Three days per week, patients attend group-based treatment for two-and-a-half hours per day. The fourth day of each week consists of a one-hour group-based treatment, a one-hour family meeting, and a one-hour exposure session that includes children and their caregivers. One day per week, parents also attend a one-hour parent guidance group as part of the overall treatment package. Patients also have psychopharmacology consultations with the program psychiatrist on a case-by-case basis. On their first birthday that falls after the date of discharge, patients are sent a birthday card that includes a greeting and reminders about coping skills that they learned in the program.

The investigators expect to recruit at least 45 assenting/consenting patients in the first year of the study. The plan is to treat six-to-eight patients during each one-month module and to have a waitlist, if interest in the program exceeds the program's capacity. If a waitlist exists, patients, who are on this waitlist, will be evaluated as the study's control group once they are four weeks away from their target admission date.

Before the patient's first assessment through the program, a clinician will inform the patient and caregivers about the opportunity to participate in a voluntary research study at the McLean Anxiety Mastery Program. Assent/consent will be requested to utilize these data for research purposes. The patient and caregivers will be told that all of the information gathered from the child- and caregiver-report measures are part of routine clinical practice, and permission is being sought to use this de-identified data for research purposes. The patient and caregivers will be reminded that their decision to or not to participate in the research study will not affect the treatment they receive.

The assessments are conducted at the following time points: 1) upon admission, 2) weekly while the patients are participating in treatment, 3) upon discharge, and 4) at a three-month follow-up visit.

The child- and parent--report questionnaires are administered through REDCap Survey, a secure, HIPAA-compliant program for building and managing online surveys. The measures are completed on families' devices at home. If a patient or family member does not complete the online survey within 48 hours, a clinician will contact them with a reminder one time via phone or e-mail. The survey does not include questions assessing risk (e.g., for suicidal ideation, self-harm, substance use).

ELIGIBILITY:
Inclusion Criteria:

* All youth who are eligible to participate in the McLean Anxiety Mastery Program will be invited to participate in the research study.
* Eligibility criteria for the McLean Anxiety Mastery Program include:

  * children and adolescents who are between the ages of 6 and 19 and
  * who present with at least one of the following disorders:

    * Separation Anxiety Disorder,
    * Social Anxiety Disorder,
    * Panic Disorder,
    * Agoraphobia,
    * Specific Phobia(s), and
    * OCD.
  * Interested and eligible patients and their caregivers should complete and submit an application (https://www.mcleanhospital.org/sites/default/files/2021-07/MAMP-Application-07032021_0.pdf) to begin the phone screen process.

Exclusion Criteria:

* Patients ineligible for the treatment program, and therefore the study, include those who have engaged in substance abuse during the six weeks prior to the first evaluation (i.e., waitlist or admission) the phone screening,
* those who report that they are unwilling to refrain from self-injurious behaviors during the waitlist and treatment periods,
* those who are experiencing active symptoms of psychosis,
* those who exhibit severe behavioral disinhibition or aggression, and
* those who express an intent and/or plan to commit suicide or homicide at the time of their first evaluation the initial phone screening.
* Patients must be fluent in English to participate in the program because all off-grounds exposure groups will be conducted in English (whenever possible, however, translation services will be provided for patients whose parents are not fluent in English).

Ages: 6 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 559 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2024-11 (Actual); Study Completion 2024-11 (Actual)

PRIMARY OUTCOMES:
Change in Score in Spence Children's Anxiety Scale (SCAS; Spence 1997). | Change between 0 weeks of treatment and after weeks of treatment, change between 4 weeks of treatment and 16 weeks after treatment
  The SCAS is a 44-item self-report inventory that measures anxiety severity.

SECONDARY OUTCOMES:
Change in Score in Center for Epidemiolgic Studies Depression Scale (CES-D; Radloff 1977). | Change between 0 weeks of treatment and after weeks of treatment, change between 4 weeks of treatment and 16 weeks after treatment
  The CES-D is a 20-item self-report inventory that measures depression severity.

OTHER OUTCOMES:
Change in Score in Spence Children's Anxiety Scale (SCAS - Parent Report; Spence 2000). | Change between 0 weeks of treatment and after weeks of treatment, change between 4 weeks of treatment and 16 weeks after treatment
  The SCAS -Parent Report is a 39-item parent report inventory that measures the child's anxiety severity.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Sperling, Ph.D., Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Cambridge, Massachusetts, United States